CLINICAL TRIAL: NCT02741154
Title: Role of Aromatase Inhibitor to Enhance Ovulation in Poor Responder During Induction With Short Antagonist Protocol in Cases of ICSI(Intracytoplasmic Sperm Injection) a Case Control Study
Brief Title: Role of Aromatase Inhibitor to Enhance Ovulation in Poor Responder During Induction With Short Antagonist Protocol in Cases of ICSI
Acronym: AIPRICSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Reham Elkhateeb, doctor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUH 20167; MUH20167 (Registry Identifier: Minia University)
Record Dates: First submitted 2016-04-12; First posted 2016-04-18 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Infertility Indicated for ICSI
Keywords: aromataze inhibitor, poor responder ,induction
MeSH Terms: interventions — Neoadjuvant Therapy; Letrozole; hMG-IBSA; ricin A-GnRH conjugate; Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aromataze group (Experimental): patients will receive induction with HMG plus aromataze inhibitor plus GnRh antagonist plus HCG injection
  Interventions: Drug: induction with aromataze inhibitor; Drug: HMG; Drug: GnRh a; Drug: HCG
- classic group (Active Comparator): same protocol for induction without aromataze inhibitor
  Interventions: Drug: HMG; Drug: GnRh a; Drug: HCG

INTERVENTIONS:
Drug: induction with aromataze inhibitor — letrozole 2.5mg once daily start in the first day of menses for 5days
  Other Names: letrozole
  Arms: aromataze group
Drug: HMG — HMG 300 IU injection once daily start at first day of menses with follow up by trans vaginal ultrasound (TVUS ) till at least three follicles reach 14 mm in diameter
  Other Names: merional
Drug: GnRh a — antagonist given 0.1 ml injection once daily with continous follow up when at least three follicles reach 17mm in diameter HCG 10.000 IU injection and ovum pick up 24-36hours after injection
  Other Names: decapeptyl
Drug: HCG — 10.000 IU HCG injection when at least three follicles reach 17mm in diameter
  Other Names: choriomon

SUMMARY:
study the effect of aromataze inhibitor induction together with short stimulation protocol by gonadotrphin releasing hormon antagonist in cases that expected to be poor responder before ICSI

DETAILED DESCRIPTION:
This is a prospective randomized case control study will be conducted in Maternity hospital IVF unite Minia University after being approved by local ethical committee of obstetrics and gynecology department faculty of medicine, all study details will be explained to patients and informed consent will be obtained before inclusion in the study . enrolled patients will be randomized into two groups using simple randomization by sealed opaque envelops contain serial computer generated numbers Control group will receive HMG 300 IU daily start at first day of menses with follow up by trans vaginal ultrasound (TVUS ) when at least three follicles reach 14mm diameter GnRh antagonist given 0.1 ml continue follow up when at least three follicles reach 17mm in diameter ovum pickup will done under TVUS guide if less than three follicles cycle will be cancelled .

Study group will receive same management plus letrozole 2.5mg daily start at the first day of menses for 5 days and continue with same protocol

ELIGIBILITY:
Inclusion Criteria:

* infertlity indicated for ICSI
* Ovarian factor
* Tubal factor
* Unexplained infertility
* poor responders

Exclusion Criteria:

* Expected high responder
* Endometriosis
* Male and uterine factors
* Ovarian mass or cyst

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08-12; Primary Completion 2017-08-24 (Actual); Study Completion 2017-09-03 (Actual)

PRIMARY OUTCOMES:
Number of follicles per cycle that reach more than 17mm in diameter(quantity of ova) | day of HCG injection
  measurement of the diameter of follicles by transvaginal ultrasoundand description of diameter in report
quality of ova | day of ovum pick up
  After ova picking up examination of all ova under microscope and report how many ova reach metaphase II (quality) if more than 3 ova reach metaphase II considered satisfactory quality of ova in the current cycle

SECONDARY OUTCOMES:
pregnancy rate | 14 days after ovum pick up
  presence of clinical pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mitwally MF, Casper RF. Aromatase inhibition improves ovarian response to follicle-stimulating hormone in poor responders. Fertil Steril. 2002 Apr;77(4):776-80. doi: 10.1016/s0015-0282(01)03280-0. PMID 11937133